CLINICAL TRIAL: NCT00762879
Title: Spine Quantitative Computed Tomography (QCT) for the Assessment of Osteoporosis on Children
Brief Title: Spine Quantitative Computed Tomography (QCT)
Acronym: Spine QCT
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: 07-005528
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: Juvenile Idiopathic Arthritis; JIA; Arthritis; Osteoporosis; Osteoporosis in Children
MeSH Terms: conditions — Arthritis, Juvenile; Arthritis; Osteoporosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment

SUMMARY:
The purpose of this study is to compare healthy children to children who have a chronic illness called Juvenile Idiopathic Arthritis (JIA). JIA is a childhood disease that causes swollen joints that are often stiff and painful. JIA affects about 1 in 1,000 children age 16 and younger.

DETAILED DESCRIPTION:
Children with chronic illnesses are at risk for bone fragility due to inflammation, glucocorticoid therapy, physical activity limitation, malnutrition, and pubertal delay. The impact of low bone mass during childhood may be immediate, resulting in childhood fractures, or delayed, due to suboptimal peak bone mass attainment.

ELIGIBILITY:
Inclusion Criteria:

* for JIA patients: subjects age 5-21 Drawn from Dr. Burnham's prospective cohort study of bone health in 101 children with arthritis.
* for Control patients: subjects age 5-21 Controls will be a 50% male/female

Exclusion Criteria:

* for JIA patients: Subjects with JIA will be excluded if they have conditions or drug exposure unrelated to JIA and known to impact growth or bone health.
* for Control patients: Chronic disease or syndrome known to affect growth or bone health, prematurity (<37 weeks gestation), or use of any medication known to affect growth.

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 200 control patients and 30 study patients
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2008-04; Primary Completion 2014-01 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Lumbar spine volumetric Bone Mineral Density (vBMD) and vertebral size will vary according to sex, age and pubertal stage. | same day

SECONDARY OUTCOMES:
Children with JIA will have lower vertebral stiffness and strength, compared with controls. | same day

CONTACTS AND LOCATIONS:
Overall Officials: Jon Burnham, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States